CLINICAL TRIAL: NCT03011385
Title: Physical Activity and Health-related Quality of Life: Dyadic Research in the Context of Forming Individual, Dyadic, and Collaborative Plans. Trial 3
Brief Title: Effects of Individual, Dyadic, and Collaborative Plans on Physical Activity in Partner-Partner Dyads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014/15/B/HS6/00923_C
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Individual Planning (Experimental): The planning materials and forms have sections: (a) information on the importance of planning, including examples of how planning works and what it affects, (b) instructions of what should be included in a good plan (the when, where, and how components), (c) formulating action and coping plans.
  Action plans (referring to when, when, and how the individual will act) as well as coping plans (referring to how to overcome potential difficulties, risky situations or temptations to not engage in physical activity) will be formed. Each participant will form their plans individually, without consulting the dyadic partner, but discussing the plans with the experimenter.
  Interventions: Behavioral: Individual Planning; Behavioral: Education
- Dyadic Planning (Experimental): The planning materials and forms have sections: (a) information on the importance of planning, including examples of how planning works and what it affects, (b) instructions of what should be included in a good plan (the when, where, and how components), (c) formulating action and coping plans.
  Action plans as well as coping plans will be formed. Both partners in the dyad jointly form one plan. This jointly developed plan is discussed with the experimenter.
  The plan focuses on physical activity of only one person in the dyad. This target person will be selected jointly by the participants if both participants are healthy. If one participant has a chronic disease, e.g. diabetes or a cardiovascular disease, the plans are formed for the person with a disease.
  Interventions: Behavioral: Dyadic Planning; Behavioral: Education
- Collaborative Planning (Experimental): The planning materials and forms have sections: (a) information on the importance of planning, including examples of how planning works and what it affects, (b) instructions of what should be included in a good plan (the when, where, and how components), (c) formulating action and coping plans.
  Action plans and coping plans will be formed. Both partners in the dyad jointly form one plan. This jointly developed plan is discussed with the experimenter.
  The plan focuses on physical activity of both persons within the dyad (both partners) and include some plans for joint physical activity.
  Interventions: Behavioral: Collaborative Planning; Behavioral: Education
- Education (Active Comparator): The education materials address physical activity and healthy nutrition guidelines for age groups and chronic disease. Participants receive a set of educational materials about types of physical activity (PA), PA intensity, exercise calorie expenditure, strength and endurance training, stretching, and general nutrition guidelines in terms of meal composition, and nutrients, meal frequency. The materials exclude any planning statements. The education is delivered by the experimenter to a partner-partner dyad and discusses individual guidelines for both dyadic partners.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Individual Planning — Participants are filling in the planning forms, referring to their individual physical activity. Both members of the dyad form their own, interdependent plans.
  The following behavior change techniques (BCT) are included in the planning intervention protocol: action planning, barrier identification, prompting self-talk, relapse prevention/coping planning. Applications of all BCT included references to planning.
  Arms: Individual Planning
Behavioral: Dyadic Planning — Participants are filling in the planning forms jointly. Planning refers to physical activity of only one person in the dyad. The other person in the dyad is actively participating in forming plans by the target person.
  The following BCT are included in the planning intervention protocol: action planning, barrier identification, prompting self-talk, relapse prevention/ coping planning. Applications of all BCT included references to planning.
  Arms: Dyadic Planning
Behavioral: Collaborative Planning — Participants are filling in the planning forms jointly. Planning refers to physical activity of both persons in the dyad. Physical activity may be performed jointly by both persons in the dyad. The following BCT are included in the planning intervention protocol: action planning, barrier identification, prompting self-talk, relapse prevention/ coping planning. Applications of all BCT included references to planning.
  Arms: Collaborative Planning
Behavioral: Education — The education group participants receive extended physical activity and healthy nutrition education program. The education includes: (1) the guidelines for physical activity and healthy nutrition, tailored to age and health status of the participants, (2) the examples of exercises and their metabolic equivalent; (3) information about healthy body mass and body composition.

SUMMARY:
OBJECTIVE: The project aims at investigating of the effects of three types of planning (individual planning, collaborative planning, and dyadic planning) on physical activity among dyads.The influence of three planning interventions are compared with an active control condition, including physical activity education.

PARTICIPANTS: The effects of the interventions are evaluated among dyads of two adults (partner-partner dyads). Adults forming dyads (e.g. two romantic partners, two relatives, two co-workers, two friends) who are in regular contact for at least one year will be enrolled. A minimum of 50 dyads enrolled into the each arm of the trial (a total of 200 dyads). The interventions consist of six planning sessions.

DESIGN: The dyads are randomly assigned to one of four experimental conditions. The assessment of the main and secondary outcomes is conducted at the baseline, at 1 week after the first intervention session, at post-intervention (after six intervention sessions are completed), and at 6-, and 12-month follow-ups.

OUTCOMES: Physical activity constitutes the main outcome, whereas health-related quality of life (HRQOL), body mass index, and sedentary behavior as well as the self-regulatory strategy called the use of planning (individual, dyadic and collaborative) are secondary outcomes.

DETAILED DESCRIPTION:
Individual planning (also known as implementation intentions or action and coping planning) is a regulatory strategy, which refers to making plans on when, where, and how to perform an intended behavior. In dyadic planning, a target person is setting plans together with a partner on when, where, and how the target person will individually engage in behavior change. The concept of dyadic planning differs from the conceptualization of collaborative plans, where two individuals make plans on how to enact a behavior together.

The study will evaluate the effects of a short-term planning intervention. The intervention includes a total of six sessions: two face-to-face sessions with the experimenter (delivered over two weeks) and three sessions delivered over phone (over the following three weeks), one face-two-face session (delivered at one month after the third session delivered over the phone). The delivery has an individual format (the experimenter + the dyad). The total time from first to sixth session is 2 months. The setting for the interventions will include physician's offices and participant's home. The same format, schedule, delivery, and setting will be used for conducting active control group procedures.

ELIGIBILITY:
Inclusion Criteria:

* Both partners in the dyad are adults
* At least one partner in the dyad does not meet the World Health Organization guidelines for physical activity for their respective age group and health status
* Participants are healthy or with a diagnosed chronic illness (without contraindications for moderate intensity physical activity
* The partners may be a romantic relationship or in another relationship: next of kin, family members, friends who are willing to join the study together
* The dyadic partners are in the stable relationship for at least one year or meet and spend time together regularly for at least one year

Exclusion Criteria:

* Any existing diseases with contraindications for moderate intensity physical activity, confirmed by patient's primary care physician or a specialist in cardiovascular diseases/endocrinology/rehabilitation medicine providing care for the patient during the recruitment and follow-ups
* Both participants in the dyad meet the World Health Organization guidelines for physical activity for their respective age group and health status in terms of minutes per week, the intensity of physical activity, and the types of exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Physical activity | Change from baseline physical activity at 8 months
  Accelerometry: ActiGraph (the model: wGT3X-B)

SECONDARY OUTCOMES:
Health-related quality of life (HRQOL) | Change from baseline HRQOL at 8 months
  WHOQOL--BREF Questionnaire (Skevington et al., 2004)
The use of planning | Change from baseline use of planning at 2 months
  The self-reported use of planning questionnaire (individual, dyadic and collaborative), based on Luszczynska (2006)
Body mass index (BMI) | Change from baseline BMI at 8 months
  Certified and standardized body weight scales (Beurer; European Union safety certificate; measurement error < 5%) and measuring rods will be used. Body mass index will be calculated using the following formula: body weight [in kg] divided by a square of body height [in meters]. Body weight will be recorded in kilograms and body height will be recorded in meters.
Physical activity | Change from the baseline physical activity at 8 months
  The International Physical Activity Questionnaire (IPAQ) (Craig et al., 2003); open-ended questions indicating the minutes and the number of occasions of physical activity behavior per week; higher scores represent better outcome

OTHER OUTCOMES:
Habitual physical activity | Change from baseline habitual physical activity at 8 months
  Self-reported habit index questionnaire for physical activity (based on Gardner et al., 2012)
Habitual sedentary behavior | Change from baseline habitual sedentary behavior at 8 months
  Self-reported habit index questionnaire for sedentary behavior (based on Gardner et al., 2012)
Sedentary behavior | Change from baseline habitual sedentary behavior at 8 months
  Accelerometry: ActiGraph (the model: wGT3X-B)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Luszczynska, PhD, Principal Investigator — SWPS University of Social Sciences and Humanities
Locations (1):
- University of Social Sciences and Humanities, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
As agreed with the funding institution (the National Science Centre, Poland) the dataset will be publicly available (for research use) not later than in 2023 at the website of the SWPS University of Social Sciences and Humanities, Wroclaw, Poland

REFERENCES:
- [Background] Burkert S, Knoll N, Luszczynska A, Gralla O. The interplay of dyadic and individual planning of pelvic-floor exercise in prostate-cancer patients following radical prostatectomy. J Behav Med. 2012 Jun;35(3):305-17. doi: 10.1007/s10865-012-9416-2. Epub 2012 Mar 28. PMID 22454228
- [Background] Prestwich A, Conner MT, Lawton RJ, Ward JK, Ayres K, McEachan RR. Randomized controlled trial of collaborative implementation intentions targeting working adults' physical activity. Health Psychol. 2012 Jul;31(4):486-95. doi: 10.1037/a0027672. Epub 2012 Apr 2. PMID 22468716
- [Background] Luszczynska A. An implementation intentions intervention, the use of a planning strategy, and physical activity after myocardial infarction. Soc Sci Med. 2006 Feb;62(4):900-8. doi: 10.1016/j.socscimed.2005.06.043. Epub 2005 Aug 10. PMID 16095786
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Hagger MS, Luszczynska A. Implementation intention and action planning interventions in health contexts: state of the research and proposals for the way forward. Appl Psychol Health Well Being. 2014 Mar;6(1):1-47. doi: 10.1111/aphw.12017. Epub 2013 Oct 8. PMID 24591064
- [Background] Sniehotta FF, Scholz U, Schwarzer R. Action plans and coping plans for physical exercise: A longitudinal intervention study in cardiac rehabilitation. Br J Health Psychol. 2006 Feb;11(Pt 1):23-37. doi: 10.1348/135910705X43804. PMID 16480553
- [Background] Burkert S, Scholz U, Gralla O, Roigas J, Knoll N. Dyadic planning of health-behavior change after prostatectomy: a randomized-controlled planning intervention. Soc Sci Med. 2011 Sep;73(5):783-92. doi: 10.1016/j.socscimed.2011.06.016. Epub 2011 Jul 12. PMID 21807446
- [Derived] Kulis E, Szczuka Z, Keller J, Banik A, Boberska M, Kruk M, Knoll N, Radtke T, Scholz U, Rhodes RE, Luszczynska A. Collaborative, dyadic, and individual planning and physical activity: A dyadic randomized controlled trial. Health Psychol. 2022 Feb;41(2):134-144. doi: 10.1037/hea0001124. Epub 2021 Dec 30. PMID 34968130
- Available data/document: Study Protocol — https://drive.google.com/file/d/1xGrVkCeXwUZbih7NuOujjlNJcWvQ4j6H/view?usp=sharing — The file includes the protocol for data collection and intervention sessions